CLINICAL TRIAL: NCT02479620
Title: LIMBO-ATX: Lower-Limb Adventitial Infusion of DexaMethasone Via Bullfrog to Reduce Occurrence of Restenosis After Atherectomy (ATX)-Based Revascularization
Brief Title: Lower-Limb Adventitial Infusion of DexaMethasone Via Bullfrog to Reduce Occurrence of Restenosis After Atherectomy (ATX)-Based Revascularization
Acronym: LIMBO-ATX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mercator MedSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIP0173
Record Dates: First submitted 2015-06-16; First posted 2015-06-24 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Chronic Limb Ischemia
MeSH Terms: interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone Delivery (Active Comparator): Up to 60 atherectomy-based revascularization procedures at up to 30 sites in the United States and Europe.
  For Subjects randomized into the Dexamethasone Delivery arm, this protocol will utilize a 4 mg/mL preparation of Dexamethasone Sodium Phosphate Injection, USP. Each milliliter of the solution contains 4.37 mg of dexamethasone sodium phosphate equivalent to 4 mg of dexamethasone phosphate or 3.33 mg of dexamethasone. The total dose of Dexamethasone Sodium Phosphate Injection, USP will be diluted by 20% prior to infusion. This will result in a final concentration of 3.2 mg dexamethasone phosphate (3.5 mg dexamethasone sodium phosphate, or 2.67 mg dexamethasone) in each milliliter of solution.
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection, USP, 4 mg/mL
- Control (No Intervention): Up to 60 atherectomy-based revascularization procedures at up to 30 sites in the United States and Europe.
  Standard endovascular revascularization therapy consisting of atherectomy with or without angioplasty and with or without stent placement. No additional drug will be given to Subjects randomized to Control.

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate Injection, USP, 4 mg/mL — Following atherecomy-based revascularization, Investigators will be unblinded to assignment and will treat only patients assigned to the treatment arm with the Bullfrog delivery of dexamethasone.
  Arms: Dexamethasone Delivery

SUMMARY:
This is a prospective, multi-center, randomized pilot study to document the effects of adventitial delivery of dexamethasone after atherectomy-based revascularizations of lesions below the knee in symptomatic patients with critical limb ischemia (CLI).

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized pilot study to document the effects of adventitial delivery of dexamethasone after atherectomy-based revascularizations of lesions below the knee in symptomatic patients with critical limb ischemia (CLI). Up to 120 patients (60 treatment and 60 control), including up to 20 Rutherford 6 patients (10 treatment and 10 control) at up to 30 sites in the United States and Europe. This study will assess the safety and effectiveness of Bullfrog Micro-Infusion Device adventitial deposition of dexamethasone in reducing inflammation and restenosis in patients with clinical evidence of chronic critical limb ischemia with an angiographically significant lesion in the infrapopliteal crural vessels.

ELIGIBILITY:
Inclusion Criteria:

Screening Criteria:

* Age ≥18 years
* Patient or patient's legal representative have been informed of the nature of the study, agrees to participate and has signed an IRB/EC approved consent form
* Female patients of childbearing potential have a negative pregnancy test ≤7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation
* Patient has documented chronic Critical Limb Ischemia (CLI) in the target limb from the popliteal artery to the ankle joint prior to the study procedure with Rutherford Category 4, 5 or 6
* Life expectancy >1 year in the Investigator's opinion

Angiographic Criteria:

* Successful revascularization of the TL with less than 30% residual stenosis, run-off down to the foot and direct in-line flow to any foot wound
* Reference vessel(s) diameter ≥2 mm
* Single or multiple atherosclerotic lesion ≥70% in at least one infrapopliteal crural target vessel including the tibioperoneal trunk that totals up to 30 cm in length (with no greater than 5 cm length of contiguous intervening normal artery), with possible extension into the popliteal artery distal to the center of the knee joint space (the P3 segment)

Exclusion Criteria:

Screening Criteria:

* Patient unwilling or unlikely to comply with visit schedule
* Planned major index limb amputation
* Active foot infection; however, osteomyelitis in the toes or mild cellulitis around the perimeter of gangrene or small ulcers are not exclusions, but osteomyelitis of the metatarsal or more proximal region would be exclusionary
* Inability to receive study medications
* Estimated glomerular filtration rate (eGFR) less than 30 mL/min, except for patients with end stage renal disease on chronic hemodialysis
* Stage 3 (per SVS WIfI classification) or worse heel ulcers or heel ulcers that are determined to be primarily neuropathic in nature

Angiographic/Procedural Criteria:

* Hemodynamically significant inflow lesion (≥50% DS) or occlusion in the ipsilateral iliac, SFA, or popliteal arteries in which there is failure to successfully treat and obtain a <30% residual stenosis
* Target lesion length is >25 cm as measured from proximal normal vessel to distal normal vessel
* Total length of lesions treated during the case (including target lesion, inflow lesions, and other non-target lesions) >25 cm
* Lesions revascularized during the index case but untreated by Bullfrog
* Use of alternative therapy, e.g. radiation therapy, as part of the index lesion treatment, or use of any drug eluting stents (DES) or drug-eluting balloon/drug-coated balloons (DEB/DCB) for treatment of any infra-inguinal lesions during the study procedure or during the initial six-month follow up period
* Previously implanted stent in the TL(s)
* Aneurysm in the target vessel
* Acute thrombus in the target limb
* Failure to cross the TL with a guide wire; however, subintimal wire crossing is allowed
* Heavy eccentric or concentric calcification at index lesion, which in the judgment of the investigator would prevent penetration of the Micro-Infusion Device needle through the vessel wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from MALE | Up to 6 Months following the procedure
  Freedom from major adverse limb event (MALE) within 6 months.
Freedom from CD-TLR | Up to 6 Months following the procedure
  Freedom from clinically driven target lesion revascularization (CD-TLR) within 6 months.
Composite clinical safety by freedom from adverse events including death, MALE, major unplanned amputation, or CD-TLR. | Up to 6 Months following the procedure
  Freedom from composite of death within 30 days from the index procedure, MALE, major unplanned amputation or CD-TLR within 6 months.
TVAL% change from post-procedure | 6 Months following the procedure
  Transverse-view vessel area loss percentage (TVAL%) of the target lesion at 6 months by quantitative vascular angiography (QVA) or prior to any CD-TLR of the target lesion before 6 months

SECONDARY OUTCOMES:
Composite clinical safety by freedom from adverse events including death, unplanned amputation, CD-TLR, SAE or MALE. | Up to 12 months following the procedure
  Freedom from composite of death, unplanned amputation and CD-TLR, serious adverse events (SAE) and MALE.
Event-free survival | 12 months following the procedure
  Proportion of patients reaching 12-month endpoint without a composite clinical safety event.
QVA change from post-procedure | 6 months following the procedure
  Improvement in % diameter stenosis (%DSS) of the target lesion (TL) and the maximum late lumen loss for the lesion (LLL) will be assessed by quantitative vascular angiography (QVA).
IVUS change from post-procedure | 6 months following the procedure
  Improvement in intravascular ultrasound (IVUS) result with in the TL (subgroup analysis).
Amputation-free survival | 30 days, 6 and 12 months following the procedure
  Percentage of patients reaching the endpoints without major or minor amputation.
Major and minor amputations and amputation level | 30 days, 6 and 12 months following the procedure
  Percentage of patients requiring amputation (major: above ankle, minor: below ankle), categorized by level on the foot, ankle, or leg.
Change in foot wounds versus baseline | 30 days, 6 and 12 Months following the procedure
  The number and total size of foot wounds, reduction in number and size of baseline wounds, and occurrence of new wounds (number and size) will be measured against baseline.
Resolved CLI death | 30 days, 6 and 12 months following the procedure
  The rate of deaths in patients who had a resolution of their critical limb ischemia (CLI).
CD-TLR | 30 days, 6 and 12 months following the procedure
Primary sustained clinical improvement versus baseline | 30 days, 6 and 12 months following the procedure
  Sustained upward shift of at least 1 category on Rutherford classification as compared to baseline without the need for repeated TLR or surgical revascularization in amputation-free surviving subjects.
Secondary sustained clinical improvement versus baseline | 30 days, 6 and 12 months following the procedure
  Sustained upward shift of at least 1 category on Rutherford classification as compared to baseline including the need for repeated TLR or surgical revascularization in amputation-free surviving subjects.
SVS WIfI score versus baseline | 30 days, 6 and 12 months following the procedure
EQ5D versus baseline | 30 days, 6 and 12 months following the procedure
Walking capacity assessment versus baseline | 30 days, 6 and 12 months following the procedure
SAE/MALE assessment | 30 days, 6 and 12 months following the procedure
Inflammatory biomarker changes from baseline | 24 hours and 30 days
Healthcare economic analysis | From baseline to 24 months
  An analysis of the economics associated with the care of patients, including number of hospital days throughout the study, return visits and hospitalizations, time from index procedure to required revascularization and number of index-lesion-related readmissions.
Infustion technical success | Intra-procedural
  The grade of distribution (A-F) around infusion sites will be used as a qualitative measure of technical success of adventitial delivery of the drug.
Revascularization success | Intra-procedural
  Establishment of antegrade flow with residual stenosis <30% by angiogram.

CONTACTS AND LOCATIONS:
Overall Officials: George Adams, MD, Principal Investigator — REX Hospital, University of North Carolina Healthcare; Donald Jacobs, MD, Principal Investigator — Saint Louis University Hospital
Locations (10):
- United States (10):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Denver Veterans Administration Hospital, Denver, Colorado
  - Mid-Michigan Heart & Vascular, Saginaw, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - St.Louis University Hospital, St Louis, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - UNC Health Care - Rex Hospital, Raleigh, North Carolina
  - Sanford Research, Sioux Falls, South Dakota
  - Tennova - Turkey Creek Medical Center, Knoxville, Tennessee
  - Mission Research Institute (New Braunfels Cardiology - GRMC), New Braunfels, Texas

IPD SHARING:
Plan to Share IPD: Yes